CLINICAL TRIAL: NCT04333199
Title: Nudging myGeisinger Enrollment Using Timely Email Messaging Reminding Patients of Lab Results Available
Brief Title: Timely Nudge About Lab Results to Increase myGeisinger Uptake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Program Director, Behavioral Insights Team, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2020-0316
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Results first posted 2021-05-03 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Telehealth; Health Behavior
Keywords: Behavioral Economics; Patient Portal
MeSH Terms: conditions — Health Behavior | interventions — Price Transparency

STUDY DESIGN:
Intervention Model Description: Every day within the designated study period, an email will be sent to patients who 1) fulfill inclusion criteria, 2) have been randomized to one of the email conditions (rather than the control group), and 3) have not already been randomized to a study condition on a previous day (i.e. no patient will be emailed for this study twice).
Who Masked: Participant
Masking Description: Participants (i.e., patients) will not be informed specifically of their assignment to different arms throughout the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Patients do not receive an email
- Timely nudge - view results (Experimental): Patients are emailed about myGeisinger when they have a lab result ready to view. The email includes a "View My Lab Results" button, which encourages them to click as a pre-commitment step that then brings them to the myGeisinger sign-up page.
  Interventions: Behavioral: Timely; Behavioral: Foot-in-the-door
- Timely nudge - get started (Experimental): Patients are emailed about myGeisinger when they have a lab result ready to view. The email includes a "Get Started With myGeisinger" button that is transparent about the next step in the process, before the patient can view test results.
  Interventions: Behavioral: Timely; Behavioral: Transparency

INTERVENTIONS:
Behavioral: Timely — Email
  Arms: Timely nudge - get started; Timely nudge - view results
Behavioral: Transparency — Email
  Arms: Timely nudge - get started
Behavioral: Foot-in-the-door — Email
  Arms: Timely nudge - view results

SUMMARY:
The purpose of the current study is to test whether sending email communications in a timely manner - when patients have laboratory results available to view on the myGeisinger patient portal - increases enrollment in the portal.

DETAILED DESCRIPTION:
Online patient portals are convenient tools that improve patient access to healthcare services while often reducing burden to both patients and providers. However, many patients have not enrolled in such portals, including Geisinger's patient portal, known as myGeisinger.

The purpose of the current study is to test whether sending myGeisinger enrollment information in a timely manner - when the benefits of enrolling are most readily available - increases enrollment. Specifically, messages will be timely in terms of lab test results having just been made available online, with the added benefit that patients can view their results prior to receiving them via mail. Unenrolled patients who recently had a laboratory procedure ordered and whose results are now ready for sharing will be informed via email that their lab results are available. At the same time, these patients will be reminded that these results can be viewed online through myGeisinger.

The primary outcome measure of interest, myGeisinger enrollment rates, will be compared between the emailed population and a control group that similarly has lab results available but will not be contacted. In addition, two different versions of the email communication will be tested. One will highlight that the patient will have to go through a sign-up process before viewing test results (in the service of transparency). The other will provide a presumed direct link to view those results, via a button that potentially serves as a pre-commitment step to undergo the registration process ("foot in the door" effect). Secondary analyses will assess differences in enrollment rates as well as unsubscribe rates between the email versions. Exploratory analyses will further examine differences in the rates at which patients opened and clicked on enrollment links within the two emails. Statistical analyses will employ generalized linear models with a binary distribution and log-link function.

ELIGIBILITY:
Inclusion Criteria:

* Geisinger patient for whom a lab was ordered within 30 days prior to email date
* Patient's lab test result released day before email date

Exclusion Criteria:

* Patient already enrolled in myGeisinger
* Patient has already declined myGeisinger

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5012 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings.
Supporting Information: Analytic Code
Time Frame: The data will become available after publication of study results in a scientific journal and will be available as long as the Open Science Framework hosts the data.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.
URL: http://osf.io

RESULTS

PARTICIPANT FLOW:
Period: Evaluated Patients
Arm/Group | Control | Timely Nudge - View Results | Timely Nudge - Get Started
Started | 1669 | 1672 | 1671
Completed (Removed patients not found in EHR) | 1669 | 1671 | 1669
Not Completed | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 2
Period: Emailed Patients
Arm/Group | Control | Timely Nudge - View Results | Timely Nudge - Get Started
Started | 0 (Patients in this group were not emailed) | 1671 | 1669
Valid Email Address (Email address not flagged as invalid by email delivery software) | 0 (Patients in this group were not emailed) | 1495 | 1441
Completed (Email delivered (did not bounce back)) | 0 (Patients in this group were not emailed) | 1399 | 1351
Not Completed | 0 | 272 | 318

BASELINE CHARACTERISTICS:
Population: Investigators did not have access to baseline demographic information for study participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Timely Nudge - View Results | Timely Nudge - Get Started | Total
Number analyzed (Participants) | 1669 | 1671 | 1669 | 5009
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Between 18 and 65 years | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  >=65 years | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Enrollment - Timely Email (Combined Email Arms) vs. no Intervention
Description: Patient enrolled in myGeisinger (yes / no)
Time Frame: 1 week post-intervention
Population: Patients who were randomized and for whom there was a record in the EHR.
Measure: Count of Participants; unit: Participants
Groups:
- Timely Nudge: Patients are emailed about myGeisinger when they have a lab result ready to view.
  Timely: Email
Arm/Group | Control | Timely Nudge
Number analyzed (Participants) | 1669 | 3340
Participants | 65 | 361
Statistical Analysis 1: Comparison: Control vs Timely Nudge; Test type: Superiority; p < 0.001, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 2.9903891, 95% CI 2-sided [2.2805876 to 3.9211066]

2. Secondary Outcome: Enrollment - Email Including a "Get Started" Button vs. a "View Results" Button
Description: Patient enrolled in myGeisinger (yes / no)
Time Frame: 1 week post-intervention
Population: Patients who were delivered an email (i.e. email did not bounce back) and for whom there was a record in the EHR.
Measure: Count of Participants; unit: Participants
Arm/Group | Timely Nudge - View Results | Timely Nudge - Get Started
Number analyzed (Participants) | 1399 | 1351
Participants | 190 | 159
Statistical Analysis 1: Comparison: Timely Nudge - View Results vs Timely Nudge - Get Started; Test type: Superiority; p = 0.154, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 1.1781659, 95% CI 2-sided [0.9404654 to 1.4759445]

3. Secondary Outcome: Email Opened - Email Including a "Get Started" Button vs. a "View Results" Button
Description: Email was opened (yes / no)
Time Frame: 1 week post-intervention
Population: Patients who were delivered an email (i.e. email did not bounce back) and for whom there was a record in the EHR.
Measure: Count of Participants; unit: Participants
Arm/Group | Timely Nudge - View Results | Timely Nudge - Get Started
Number analyzed (Participants) | 1399 | 1351
Participants | 654 | 617
Statistical Analysis 1: Comparison: Timely Nudge - View Results vs Timely Nudge - Get Started; Test type: Superiority; p = 0.571, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 0.9575636, 95% CI 2-sided [0.8242111 to 1.1124918]

4. Secondary Outcome: Link Clicked - Email Including a "Get Started" Button vs. a "View Results" Button
Description: Link / button to start the enrollment process was clicked (yes / no)
Time Frame: 1 week post-intervention
Population: Patients who were delivered an email (i.e. email did not bounce back) and for whom there was a record in the EHR.
Measure: Count of Participants; unit: Participants
Arm/Group | Timely Nudge - View Results | Timely Nudge - Get Started
Number analyzed (Participants) | 1399 | 1351
Participants | 494 | 307
Statistical Analysis 1: Comparison: Timely Nudge - View Results vs Timely Nudge - Get Started; Test type: Superiority; p < 0.001, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 1.8562672, 95% CI 2-sided [1.5692523 to 2.1957769]

5. Secondary Outcome: Unsubscribed - Email Including a "Get Started" Button vs. a "View Results" Button
Description: Patient unsubscribed from these email communications (yes / no)
Time Frame: 1 month post-intervention
Population: Patients who were delivered an email (i.e. email did not bounce back) and for whom there was a record in the EHR.
Measure: Count of Participants; unit: Participants
Arm/Group | Timely Nudge - View Results | Timely Nudge - Get Started
Number analyzed (Participants) | 1399 | 1351
Participants | 2 | 2

6. Secondary Outcome: Enrollment - Timely Email (Combined Email Arms) vs. no Intervention
Description: Patient enrolled in myGeisinger (yes / no)
Time Frame: 1 month post-intervention
Population: Patients who were randomized and for whom there was a record in the EHR.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Timely Nudge
Number analyzed (Participants) | 1669 | 3340
Participants | 141 | 488
Statistical Analysis 1: Comparison: Control vs Timely Nudge; Test type: Superiority; p < 0.001, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 1.8542767, 95% CI 2-sided [1.5220654 to 2.2589975]

ADVERSE EVENTS:
Time Frame: No adverse events were evaluated.
Description: We only received information about email engagement and portal enrollment. We did not collect or receive any information regarding adverse events.
Arm/Group | Control | Timely Nudge - View Results | Timely Nudge - Get Started
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
For this study, we only received data about engagement with the email and enrollment in the patient portal. Demographic information such as age, sex, or gender were not collected. Note that for some patients, enrollment data could not be extracted from Geisinger's electronic health records; these patients were excluded from analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT04333199/Prot_SAP_000.pdf